CLINICAL TRIAL: NCT03465865
Title: Visual Acuity and Optical Coherence Tomography One Year After ILM-flap Transposition for Surgical Repair of Macular Holes
Brief Title: Visual Acuity and Optical Coherence Tomography One Year After ILM-flap Transposition
Status: Completed | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, head of the department of ophthalmology, professor, MBA, Vienna Institute for Research in Ocular Surgery
Other Study IDs: ILMflap
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Macular Hole
MeSH Terms: conditions — Retinal Perforations | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- ILM-flap: Patients after surgical repair of macular holes with ILM-flap transposition are invitied to a follow-up for optical coherence tomography and visual acuity testing one year after surgery
  Interventions: Device: optical coherence tomography

INTERVENTIONS:
Device: optical coherence tomography — optical coherence tomography enables diagosis of macular structures and therefore provides information on macular hole closure.
  Other Names: visual acuity test

SUMMARY:
ILM-flap (internal limiting Membrane-flap) transposition is a new surgical option in repair of macular holes, therefore one year outcomes are needed to better evaluate that method.

DETAILED DESCRIPTION:
Patients that have been scheduled for vitrectomy with ILM-flap transposition, a new surgical option in repair of macular holes, are invited to a follow-up one year after surgery, including optical coherence tomography and visual acuity testing.

ELIGIBILITY:
Inclusion Criteria:

* history of ILM-flap transposition

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are invited for a follow-up one year after ILM-flap transposition for surgical repair of macular holes
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
OCT | 5 minutes
  macular hole closure is assessed with optical coherence tomography

SECONDARY OUTCOMES:
visual acuity | 5 minutes
  visual acuity describes functional outcomes of the eye

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof, Principal Investigator — VIROS at Hanuschkrankenhaus Vienna
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No